CLINICAL TRIAL: NCT05081492
Title: A Phase I, First-in-Human Study of Intratumoral Administration of CF33-hNIS-antiPDL1, A Novel Chimeric Oncolytic Poxvirus Encoding Human Sodium Iodide Symporter (HNIS) in Patients With Metastatic Triple Negative Breast Cancer
Brief Title: CF33-hNIS-antiPDL1 for the Treatment of Metastatic Triple Negative Breast Cancer
Status: Active, not recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: City of Hope Medical Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH); Imugene Limited (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 21094; NCI-2021-08983 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); 21094 (Other: City of Hope Medical Center); P30CA033572 (NIH)
Record Dates: First submitted 2021-10-04; First posted 2021-10-18 (Actual); Last update posted 2025-10-06 (Actual); Status verified 2025-10

CONDITIONS: Anatomic Stage IV Breast Cancer AJCC v8; Metastatic Triple-Negative Breast Carcinoma; Prognostic Stage IV Breast Cancer AJCC v8
MeSH Terms: conditions — Triple Negative Breast Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- Treatment (CF33-hNIS-antiPDL1) (Experimental): Patients receive CF33-hNIS-antiPDL1 IT on days 1 and 15. Treatment repeats every 28 days for up to 3 cycles in the absence of disease progression or unacceptable toxicity.
  Interventions: Biological: Oncolytic Virus CF33-expressing hNIS/Anti-PD-L1 Antibody

INTERVENTIONS:
Biological: Oncolytic Virus CF33-expressing hNIS/Anti-PD-L1 Antibody — Given IT
  Other Names: CF33 Expressing hNIS-Anti-PD-L1 Antibody; CF33-hNIS-antiPDL1

SUMMARY:
This phase I trial tests the safety, side effects, and best dose of CF33-hNIS-antiPDL1 in treating patients with triple negative breast cancer that has spread to other places in the body (metastatic). CF33-hNIS-antiPDL1 is an oncolytic virus. This is a virus that is designed to infect tumor cells and break them down.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVE:

I. To determine the safety and tolerability of a novel chimeric oncolytic orthopoxvirus, oncolytic virus CF33-expressing hNIS/Anti-PD-L1 antibody (CF33-hNIS-antiPDL1), by the evaluation of toxicities including: type, frequency, severity, attribution, time course, reversibility and duration according to Common Terminology Criteria for Adverse Events (CTCAE) 5.0 criteria.

SECONDARY OBJECTIVES:

I. To determine the optimal biologic dose (OBD) (defined as a safe dose that induces an immune response in tumors [increase checkpoint target PD-L1 by at least 5% and/or increase T cell infiltration by at least 10%]) and the recommended phase II dose (RP2D) for future expansion trial.

II. To determine tumor response rates by Response Evaluation Criteria in Solid Tumors (RECIST) version (v)1.1 (primary) and immune-modified (i)RECIST (secondary).

III. To document possible therapeutic efficacy and evaluate progression-free survival, overall survival and response.

EXPLORATORY OBJECTIVE:

I. To determine the immune and genomic profiles of tumors before and after CF33-hNIS-antiPDL1 therapy.

OUTLINE: This is a dose-escalation study.

Patients receive CF33-hNIS-antiPDL1 intratumorally (IT) on days 1 and 15. Treatment repeats every 28 days for up to 3 cycles in the absence of disease progression or unacceptable toxicity.

After completion of study treatment, patients are followed up at 30 days, then every 3 months for 1 year.

ELIGIBILITY:
Inclusion Criteria:

* Documented informed consent of the participant and/or legally authorized representative

  * Assent, when appropriate, will be obtained per institutional guidelines
* Agreement to research biopsies on study, once during study and end of study, exceptions may be granted with study principal investigator (PI) approval
* >= 18 years
* Eastern Cooperative Oncology Group (ECOG) =< 2
* Histologically confirmed metastatic triple negative breast cancer. Triple negative status will be defined as estrogen receptor (ER) and progesterone receptor (PR) =< 10% by immunohistochemistry (IHC) and HER2 negative, per American Society of Clinical Oncology/College of American Pathologists (ASCO/CAP) guidelines
* Measurable disease by RECIST 1.1
* Patients must have progressed on or been intolerant of at least 2 prior lines of therapy for advanced/metastatic disease. Patients that qualify for immunotherapy and/or PARP inhibitors must have progressed on or been intolerant of these agents
* Fully recovered from the acute toxic effects (except alopecia) to =< grade 2 to prior anti-cancer therapy
* Must have a superficial tumor (cutaneous, subcutaneous), breast lesion or nodal metastases amenable to safe repeated intratumoral injections per treating physician and interventional radiologist review
* Absolute neutrophil count (ANC) >= 1,500/mm^3

  * NOTE: Growth factor is not permitted within 14 days of ANC assessment unless cytopenia is secondary to disease involvement
* Platelets >= 100,000/mm^3

  * NOTE: Platelet transfusions are not permitted within 14 days of platelet assessment unless cytopenia is secondary to disease involvement
* Total bilirubin =< 1.5 X upper limit of normal (ULN)
* Aspartate aminotransferase (AST) =< 2.5 x ULN

  * If liver metastases are present: AST =< 5 x ULN
* Alanine aminotransferase (ALT) =< 2.5 x ULN

  * If liver metastases are present: ALT =< 5 x ULN
* Serum creatinine =< 1.5 mg/dL or creatinine clearance of >= 50 mL/min per 24 hour urine test or the Cockcroft-Gault formula
* Prothrombin (PT) =< 1.5 x ULN
* Activated partial thromboplastin time (aPTT) =< 1.5 x ULN
* Women of childbearing potential (WOCBP): negative serum pregnancy test
* Agreement by females and males of childbearing potential* and their partners to use an effective method of birth control (defined as a hormonal or barrier method) or abstain from heterosexual activity for the course of the study through at least 6 months after the last dose of protocol therapy

  * Childbearing potential defined as not being surgically sterilized (men and women) or have not been free from menses for > 1 year (women only)

Exclusion Criteria:

* Chemotherapy, biological therapy, immunotherapy or investigational therapy within 14 days prior to day 1 of protocol therapy
* Major surgery or radiation therapy within 28 days of study therapy
* Has received a vaccination within 30 days of first study injection
* History of allergic reactions attributed to compounds of similar chemical or biologic composition to study agent
* Clinically significant uncontrolled illness
* Active infection requiring antibiotics
* Known history of immunodeficiency virus (HIV)
* Patients with a known history of hepatitis B or hepatitis C infection who have active disease as evidenced by hepatitis (Hep) B surface antigen status or Hep C polymerase chain reaction (PCR) status obtained within 14 days of cycle 1, day 1
* Another malignancy within 3 years, except non-melanomatous skin cancer
* Females only: Pregnant or breastfeeding
* Patients may not have clinically unstable brain metastases. Patients may be enrolled with a history of treated brain metastases that are clinically stable for >= 4 weeks prior to start of study treatment
* Any other condition that would, in the Investigator's judgment, contraindicate the patient's participation in the clinical study due to safety concerns with clinical study procedures
* Prospective participants who, in the opinion of the investigator, may not be able to comply with all study procedures (including compliance issues related to feasibility/logistics)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 9 (Actual)
Dates: Start 2021-10-18 (Actual); Primary Completion 2026-03-30 (Estimated); Study Completion 2026-03-30 (Estimated)

PRIMARY OUTCOMES:
Incidence of adverse events | Up to 30 days
  Toxicity will be graded according to the National Cancer Institute-Common Terminology Criteria for Adverse Events version 5.0. Observed toxicities/adverse events will be summarized in terms of type (organ affected or laboratory determination), severity, time of onset, duration, probable association with the study treatment and reversibility or outcome.

SECONDARY OUTCOMES:
Immune Biomarker Expression | Up to 6 months
  Changes (%) in PD1 expression compared to baseline by immunohistochemistry
  Changes (%) in PD-L1 expression compared to baseline by immunohistochemistry
  Changes (%) CTLA-4 expression compared to baseline by immunohistochemistry
  Changes (%) CD8 cell quantification compared to baseline by Immunohistochemistry
Optimal biologic dose | Up to 3 months
  Defined as safe dose that induces an immune response in tumors (increase checkpoint target PD-L1 by at least 5% and/or increase T cell infiltration by at least 10%).
Response rate based on Response Evaluation Criteria in Solid Tumors (RECIST) 1.1 | Up to 6 months
  Will estimate the response rate by the percent of evaluable patients and its 95% confidence interval (C.I.) by the exact method.
Response rate based on immune related iRECIST | Up to 6 months
  Will estimate the response rate by the percent of evaluable patients and its 95% C.I. by the exact method.
Progression free survival | Up to 1 year
  Will be estimated using the Kaplan-Meier product-limit method.
Clinical benefit rate | Up to 6 months
  Percentage of patients who achieved Partial Response/ Complete Response/ Stable disease at 6 months
Event-free survival | Up to 3 years
  Event-free survival (EFS): defined as the duration of time from start of protocol treatment to time of disease relapse/progression or death due to any cause, whichever occurs earlier.
Duration of response | Up to 3 years
  Duration of response (DOR): defined as the time from the first achievement of PR and CR to time of PD.
Overall survival | Up to 3 years
  Will be estimated using the Kaplan-Meier product-limit method.

CONTACTS AND LOCATIONS:
Overall Officials: Jamie Rand, Principal Investigator — City of Hope Medical Center
Locations (1):
- City of Hope Medical Center, Duarte, California, United States

REFERENCES:
- [Derived] Rand J, Yamauchi D, Chaurasiya S, Zhang J, Deshpande S, Chong L, Seiz A, Meisen H, Fong Y, Yuan Y. hNIS-based imaging to monitor treatment with the novel oncolytic virus CF33-hNIS-antiPDL1 in humans with advanced triple negative breast cancer. Front Oncol. 2025 Aug 25;15:1565244. doi: 10.3389/fonc.2025.1565244. eCollection 2025. PMID 40933893
- [Derived] Yuan Y, Egelston C, Colunga Flores O, Chaurasiya S, Lin D, Chang H, Chong LMO, Seiz A, Shah M, Meisen WH, Tang A, Martinez N, Pickett W, Murga M, Yost SE, Stewart D, Zhang J, Ede N, Modi B, Kessler J, Rand J, Fong Y. CF33-hNIS-anti-PD-L1 oncolytic virus followed by trastuzumab-deruxtecan in a patient with metastatic triple negative breast cancer: a case study. Ther Adv Med Oncol. 2023 Nov 10;15:17588359231210675. doi: 10.1177/17588359231210675. eCollection 2023. PMID 38028143